CLINICAL TRIAL: NCT01042730
Title: Randomized Evaluation of Aggressive or Moderate Lipid Lowering Therapy With Pitavastatin in Coronary Artery Disease (REAL-CAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juntendo University (Other)
Collaborators: Tokyo University (Other); Yamaguchi University Hospital (Other); Tohoku University (Other); Kyoto University (Other); Kumamoto University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSP-LD-09
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease
Keywords: Pitavastatin; Coronary Artery Disease; Cardiovascular Disease
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitavastatin 1 mg daily (Active Comparator)
  Interventions: Drug: Pitavastatin 1 mg daily or 4 mg daily
- Pitavastatin 4 mg daily (Active Comparator)
  Interventions: Drug: Pitavastatin 1 mg daily or 4 mg daily

INTERVENTIONS:
Drug: Pitavastatin 1 mg daily or 4 mg daily — Patients who met all inclusion criteria and did not meet exclusion criteria (1) are entered in run-in period, loading pitavastatin 1 mg/day for more than 1 month when informed consent was given. (Primary registration) After 1 month, patients who did not meet exclusion criteria(2) are randomized to take pitavastatin 1 mg/day or 4 mg/day.
  Other Names: LIVALO Tablet

SUMMARY:
The purpose of this study is to evaluate the prevention of cardiovascular disease by moderate cholesterol lowering therapy, pitavastatin 1mg/day or aggressive cholesterol lowering therapy, pitavastatin 4mg/day in patients with stable coronary artery disease.

DETAILED DESCRIPTION:
It was already demonstrated by previous clinical trials that statins lower the incidence of death and cardiovascular events in patients with coronary artery disease. However, whether aggressive cholesterol lowering therapy, using high dosage of statins, is more effective than moderate cholesterol lowering therapy for the prevention of cardiovascular events in patients with coronary artery disease has not been studied in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met following all criteria are entered in run-in period, loading pitavastatin 1 mg/day for more than 1 month when informed consent was given. (Primary registration)
* Coronary artery disease patients meeting one of the following events

  * History of Acute Coronary Syndrome (AMI or Unstable angina)
  * History of revascularization (PCI or CABG)
  * Diagnosis of ischemic heart disease and coronary artery stenosis as having 75% or higher stenosis according to the AHA classification
* Hypercholesterolemia patients meeting one of following criteria

  * LDL-C is 140 mg/dL or over
  * LDL-C is 100 mg/dL or over and requiring cholesterol lowering drugs judged by attending physicians
  * Patents receiving cholesterol lowering drugs
* Age (≧20 <80 year-old)
* Patients given written informed consent.

Exclusion Criteria:

Exclusion Criteria(Pre-Run-in period)

* Patients planning revascularization
* Malignant tumor in active phase
* Patients who meet contraindication of LIVALO tablet below

  * Patients who have hypersensitivity to LIVALO tablet
  * Patients who have severe liver dysfunction or biliary atresia
  * Patients who are being treated with cyclosporine
  * Pregnant women, women suspected of being pregnant, or lactating women
* Patients who have heart failure NYHA III or greater
* Patients undergoing dialysis
* Patients with familial hypercholesterolemia
* Patients registered in the other clinical trials
* Patients taking prohibited drugs
* Patients who are ineligible in the opinion of the investigator

Exclusion Criteria(Post-Run-in period)

* LDL-C is 120mg/dL or over after Run-in period
* Patients with occurrence of acute coronary syndrome (AMI or Unstable angina) within 3 months
* Patients who have been undergone PCI or CABG within 3 months
* Compliance is less than 50% in Run-in period
* Patients who met primary endpoint in Run-in period.
* Patients who met adverse events in Run-in period and judged as ineligible in the opinion of the investigator
* Patients who are ineligible in the opinion of the investigator

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13054 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of one of following events(Cardiovascular death, Non-fatal Myocardial Infarction (MI), Non-fatal Cerebral Infarction (CI), Unstable angina requiring urgent hospitalization) | 3-6 years

SECONDARY OUTCOMES:
Composite cardiovascular events | 3-6 years
Composite coronary heart disease events | 3-6 years
Composite cerebrovascular events | 3-6 years
Death events | 3-6 years
Heart disease events | 3-6 years
Cerebrovascular events | 3-6 years
The other events | 3-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Ryozo Nagai, MD, PhD, Principal Investigator — Department of Cardiovascular Medicine, University of Tokyo Graduate School of Medicine; Masunori Matsuzaki, MD, PhD, Principal Investigator — Division of Cardiology, Department of Medicine and Clinical Science, Yamaguchi University Graduate School of Medicine
Locations (2):
- Japan (2):
  - Kyoto University Hospital, Kyoto
  - Juntendo University School of Medicine, Tokyo

REFERENCES:
- [Derived] Yoshiki Y, Ozaki Y, Abe M, Ismail TF, Takahashi H, Akao M, Kawai H, Muramatsu T, Harada M, Ohta M, Hashimoto Y, Shiki Y, Koshikawa M, Miyajima K, Takatsu H, Niwa Y, Kawashima N, Ozaki R, Tsuboi N, Iimuro S, Iwata H, Sakuma I, Nakagawa Y, Hibi K, Hiro T, Fukumoto Y, Hokimoto S, Miyauchi K, Ogawa H, Daida H, Shimokawa H, Izawa H, Kimura T, Nagai R; REAL-CAD investigators. Influence of Worsening Renal Function and Baseline Chronic Kidney Disease on Clinical Outcomes in Patients With Chronic Coronary Syndromes: Insights From the REAL-CAD Study. J Am Heart Assoc. 2025 Jan 21;14(2):e034627. doi: 10.1161/JAHA.124.034627. Epub 2025 Jan 17. PMID 39818975
- [Derived] Iwata H, Miyauchi K, Naito R, Iimuro S, Ozaki Y, Sakuma I, Nakagawa Y, Hibi K, Hiro T, Fukumoto Y, Hokimoto S, Saito Y, Ogawa H, Shimokawa H, Daida H, Kimura T, Nagai R. Significance of Persistent Inflammation in Patients With Chronic Coronary Syndrome: Insights From the REAL-CAD Study. JACC Adv. 2024 Jun 5;3(7):100996. doi: 10.1016/j.jacadv.2024.100996. eCollection 2024 Jul. PMID 39130048
- [Derived] Sakuma M, Iimuro S, Shinozaki T, Kimura T, Nakagawa Y, Ozaki Y, Iwata H, Miyauchi K, Daida H, Suwa S, Sakuma I, Nishihata Y, Saito Y, Ogawa H, Matsuzaki M, Ohashi Y, Taguchi I, Toyoda S, Inoue T, Nagai R. Optimal target of LDL cholesterol level for statin treatment: challenges to monotonic relationship with cardiovascular events. BMC Med. 2022 Nov 14;20(1):441. doi: 10.1186/s12916-022-02633-5. PMID 36372869
- [Derived] Taguchi I, Iimuro S, Iwata H, Takashima H, Abe M, Amiya E, Ogawa T, Ozaki Y, Sakuma I, Nakagawa Y, Hibi K, Hiro T, Fukumoto Y, Hokimoto S, Miyauchi K, Yamazaki T, Ito H, Otsuji Y, Kimura K, Takahashi J, Hirayama A, Yokoi H, Kitagawa K, Urabe T, Okada Y, Terayama Y, Toyoda K, Nagao T, Matsumoto M, Ohashi Y, Kaneko T, Fujita R, Ohtsu H, Ogawa H, Daida H, Shimokawa H, Saito Y, Kimura T, Inoue T, Matsuzaki M, Nagai R. High-Dose Versus Low-Dose Pitavastatin in Japanese Patients With Stable Coronary Artery Disease (REAL-CAD): A Randomized Superiority Trial. Circulation. 2018 May 8;137(19):1997-2009. doi: 10.1161/CIRCULATIONAHA.117.032615. PMID 29735587